CLINICAL TRIAL: NCT04148053
Title: Evaluation of TB-antigen Responsive T Cell Markers in Diagnosis of Tuberculosis and Extrapulmonary Tuberculosis
Brief Title: Evaluation of Immune Cell Markers in Diagnosis of Tuberculosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Caicun Zhou, Director, Department of Thoracic Oncology, Tongji University
Other Study IDs: CTB18001
Record Dates: First submitted 2019-10-29; First posted 2019-11-01 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Tuberculosis Infection
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Active TB: Subjects met the following:
  1. Either Pulmonary or Extra-pulmonary tuberculosis patients
  2. TB Bacteriological evidence obtained by culture or Xpert MTB/RIF from at least 1 specimen.
  Interventions: Diagnostic Test: TB-antigen responsive T cell markers
- Latent TB: Subjects met the following:
  1. TB Contact in history.
  2. Chest X-ray suggestive of non-TB.
  3. without any symptoms suggestive of TB.
  4. TST and/or IGRA positive.
  Interventions: Diagnostic Test: TB-antigen responsive T cell markers

INTERVENTIONS:
Diagnostic Test: TB-antigen responsive T cell markers — A blood test including a series of T cell markers which are responsive to TB antigens

SUMMARY:
Diagnosis of active and latent pulmonary tuberculosis, as well as extrapulmonary tuberculosis, is still a major challenge of TB control in China. This observational study aims to evaluate TB-antigen responsive T cell markers in the diagnosis of tuberculosis and extrapulmonary tuberculosis and try to find new prompt and cost-effective laboratory tests for active TB screening.

DETAILED DESCRIPTION:
The enrolled patients will be grouped into active or latent tuberculosis according to the bacteriological evidence of TB. The TB-antigen responsive T cell markers will be examined. The performance of each T cell marker for the diagnosis of active TB will be systematically evaluated.

ELIGIBILITY:
Inclusion Criteria:

* any patients suspicious of TB infection
* TB culture and Xpert test required
* Chest X-ray required

Exclusion Criteria:

* anti-TB therapy before the sample collection.

Ages: 7 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Any patients suspicious of TB infection
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-03-01 (Estimated)

PRIMARY OUTCOMES:
Positive rate and negative rate | 2-3 month after sampling
  Evaluation of the positive rate and negative rate for each T cell marker
Receiver operating characteristic curve | 2-3 month after sampling
  The AUC of each T cell marker will be analyzed and compared

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data will be decided by the sponsor after the accomplishment of the study.